CLINICAL TRIAL: NCT02254928
Title: Comparative Study Between the Use of Corifollitropin Alfa and Daily Recombinant FSH in the Controlled Ovarian Stimulation of Poor Responders
Brief Title: Corifollitropin Alfa Versus Daily rFSH in the Controlled Ovarian Stimulation of Poor Responders
Acronym: MANCOR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Vida Recoletas Sevilla (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other); IVI Madrid (Other); IVI Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MANCOR
Record Dates: First submitted 2014-09-25; First posted 2014-10-02 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Infertility
Keywords: poor ovarian response; controlled ovarian stimulation; randomised clinical trial; corifollitropin alfa; recombinant follicle-stimulating hormone (rFSH); human menopausal gonadotropin (HMG)
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide

ARMS (2):
- Group 1 (Other): First stimulation cycle with corifollitropin alfa (experimental) Second stimulation cycle with rFSH and HMG (active comparator)
  Interventions: Drug: Corifollitropin alfa
- Group 2 (Other): First stimulation cycle with rFSH and HMG (active comparator) Second stimulation cycle with corifollitropin alfa (experimental)
  Interventions: Drug: Corifollitropin alfa

INTERVENTIONS:
Drug: Corifollitropin alfa — One dose of 150 μg of corifollitropin alfa will be administered at day 1 of stimulation. Stimulation will be continued with 250-300 IU/day of rFSH from day 8 forward.
  Other Names: Elonva

SUMMARY:
A randomised, crossover, multicentre, national, clinical trial comparing the efficacy of corifollitropin alfa versus daily recombinant FSH and HMG in the controlled ovarian stimulation of women with a poor ovarian response undergoing IVF treatments. The main objective of this study is comparing the number of oocytes obtained after the follicle puncture when using each of these two stimulation protocols. Only poor responders according to the Bologna criteria will be recruited for this trial. All participants will undergo two stimulation cycles to obtain and accumulate oocytes by vitrification. One of the cycles will be done with the corifollitropin alfa protocol and the other with daily rFSH and HMG, the order of application of these protocols will be randomised (crossover clinical trial) in each patient.

ELIGIBILITY:
Inclusion Criteria:

* Advanced maternal age (≥40 years)
* A previous poor ovarian response (≤3 oocytes with a conventional stimulation protocol)
* An abnormal ovarian reserve test (i.e. antral follicle count <5-7 follicles or anti-mullerian hormone level <0.5-1.1 ng/ml)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of mature oocytes (metaphase II) | 1 year
  Number of mature oocytes (metaphase II) obtained after the follicle puncture

SECONDARY OUTCOMES:
Total number of oocytes | 1 year
  Total number of oocytes obtained after the follicle puncture
Symptoms associated with the ovarian stimulation protocol | 1 year
  Patients will evaluate their symptoms using a questionnaire. They will score the intensity (from 1 to 10) of each of the following symptoms: pelvic pain, headache, mood swings, nausea, tiredness, breast pain.
Patient perception of the stimulation treatment | 1 year
  Patients will evaluate how they have perceived the stimulation treatment using a questionnaire. They will score their comfort (from 1 to 10) with the following aspects of the treatment: treatment administration, number of injections and treatment length.
Length of the stimulation treatment | 1 year
  Days of stimulation treatment
Number of subcutaneous injections | 1 year
  Number of subcutaneous injections of gonadotropins (corifollitropin alfa, rFSH and HMG)

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - IVI Barcelona, Barcelona, Barcelona
  - IVI Madrid, Madrid, Madrid
  - IVI Sevilla, Seville, Seville
  - IVI Valencia, Valencia, Valencia